CLINICAL TRIAL: NCT02172404
Title: A Single-blind Two-centre Trial to Compare Administration Technique, Learning Retention of the Administration Technique and Ease of Use of the HandiHaler® With Those of the Pressurised Metered Dose Inhaler (MDI) in Patients With COPD.
Brief Title: HandiHaler® vs. Metered Dose Inhaler (MDI) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 205.220
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- HandiHaler® vs. MDI (Experimental): sequence during treatment phase: first Placebo capsule administered via HandiHaler then Ipratropium metered dose inhaler
  Interventions: Device: Placebo capsule administered via the HandiHaler®; Device: Ipratropium metered dose inhaler (MDI)
- MDI vs. HandiHaler® (Experimental): sequence during treatment phase: first Ipratropium metered dose inhaler then Placebo capsule administered via HandiHaler Ipratropium metered dose inhaler
  Interventions: Device: Placebo capsule administered via the HandiHaler®; Device: Ipratropium metered dose inhaler (MDI)

INTERVENTIONS:
Device: Placebo capsule administered via the HandiHaler®
Device: Ipratropium metered dose inhaler (MDI)

SUMMARY:
Trial to compare the administration technique for HandiHaler® vs. MDI, to compare the learning retention of the administration technique for the HandiHaler® vs. MDI and to compare the ease of use for HandiHaler® vs. MDI

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

  * Historical data (not older than 6 months) of stable airway obstruction with an forced expiratory volume at one second (FEV1) ≤ 80% of predicted normal and FEV1 ≤ 70% of forced vital capacity (FVC)
* Male or female patients with 40 years of age or older
* Smokers or ex-smokers with a smoking history of more than 10 pack-years
* Currently using a prescription bronchodilator (such as Atrovent®, Berodual®, Combivent®, salbutamol, etc.) administered at least once daily
* Able to read and understand written instructions, understand verbal instructions and fill out written questionnaires regarding the devices
* Able to give informed consent prior to participation in the trial, including discontinuation of any medications, sign an approved consent form, and be willing and able to complete all trial procedures

Exclusion Criteria:

* Any acute or chronic illness which could interfere with the conduct of completion of the trial, including but not limited to cardiovascular, renal, neurologic, liver, immunologic, or endocrine dysfunction if clinically significant
* Current or recent (past 2 years) history of drug or alcohol abuse
* Participation in any other clinical trial or use if any investigational drug within the last 30 days prior to visit 1
* Experience with the HandiHaler®
* Discontinued use of regularly prescribed use of MDI within the last 12 months.
* Treatment with any oral or injectable β-blockers within the recent 4 weeks prior to visit 1
* Treatment with oral β-adrenergics within the recent 4 weeks prior to visit 1
* Current or recent (last 6 weeks prior to visit 1) respiratory illness including, but not limited to upper or lower respiratory tract infections or asthma
* Patients who are in a pulmonary rehabilitation program or who had completed a pulmonary rehabilitation program in the 6 weeks prior to visit 1
* Patients with known hypersensitivity to ipratropium bromide, lactose or any other components of the inhalation capsule delivery system
* Patients with known sensitivity to inhaled β-agonists
* Patient using oral corticosteroid medication at unstable doses (i.e., less than 6 weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisolone per day or 20 mg every other day
* Pregnant or nursing women or women of childbearing potential not using medically approved means of contraception

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2000-10; Primary Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Performance score based on the checklist for each device | Day 0 and 28

SECONDARY OUTCOMES:
Number of errors on all scoring attempts per device use | Day 0
Number of scoring attempts per device use | Day 0
Number of incorrect answers to the "knowledge of use" questionnaire per device use | Day 28
Set of patient responses to the "ease of use" questionnaire | Day 28
Patients responses to the questionnaire | Day 28